CLINICAL TRIAL: NCT01062620
Title: A Dose Escalating Phase Ia-b Clinical Trial of the IGF-1 Receptor Inhibitor AXL1717 in Patients With Advanced Cancer: A Prospective, Single Armed, Open Label, Dose-finding Phase Ia-b Study
Brief Title: A Dose Escalating Clinical Trial of the IGF-1 Receptor Inhibitor AXL1717 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Axelar AB (Industry)
Responsible Party: Michael Bergqvist, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AXL-001
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Solid Tumors
MeSH Terms: interventions — picropodophyllin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AXL1717 (Experimental)
  Interventions: Drug: AXL1717

INTERVENTIONS:
Drug: AXL1717 — Phase I study with increasing dosage and treatment duration

SUMMARY:
A dose escalating phase Ia-b clinical trial of the IGF-1 receptor inhibitor AXL1717 in patients with advanced cancer.

The objective is to study the safety and pharmacokinetics of AXL1717 and to define an appropriate Phase 2 dose for further studies. This is the first study in man. The study is not designed to show tumor response.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Histologically confirmed diagnosis of advanced solid or haematological malignancy not amenable to standard treatment.
3. Pharmacological treatment attempt justified
4. Preserved major organ functions, i.e:

   * B-Leukocyte count ≥ 3.0 x 109/L
   * B-Neutrophil count ≥ 1.5 x 109/L
   * B-Platelet count ≥ 75 x109/L
   * B-Haemoglobin ≥ 100 g/L (transfusions are allowed)
   * P-Total bilirubin level ≤ 1.5 times the upper institutional limit of the "normal" (i.e. reference) range
   * P-ASAT or P-ALAT ≤ 2.5 times upper institutional limit of the "normal" range, ≤5 times if liver metastases have been documented
   * P-Creatinine ≤ 1.5 times upper institutional limit of the "normal" range
5. Females of childbearing potential should use adequate contraception (oral or injectable contraceptives, hormone releasing intrauterine device) throughout the study period.
6. Signed written informed consent.

Exclusion Criteria:

1. Ongoing infection or other major recent or ongoing disease that, according to the investigator, poses an unacceptable risk to the patient
2. Known malignancy in CNS
3. Prior anti-tumour therapy within 4 weeks from enrolment (6 weeks for nitrosurea and MitC).
4. Pregnancy or lactation
5. Current participation in any other interventional clinical trial
6. Performance status > ECOG 2 after optimization of analgesics
7. Life expectancy less than 3 months
8. Contraindications to the investigational product, e.g. known or suspected hypersensitivity.
9. Lack of suitability for participation in the trial, for any reason, as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-04; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To define and confirm recommended Phase 2 dose

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bergqvist, MD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Ekman S, Harmenberg J, Frodin JE, Bergstrom S, Wassberg C, Eksborg S, Larsson O, Axelson M, Jerling M, Abrahmsen L, Hedlund A, Alvfors C, Stahl B, Bergqvist M. A novel oral insulin-like growth factor-1 receptor pathway modulator and its implications for patients with non-small cell lung carcinoma: A phase I clinical trial. Acta Oncol. 2016;55(2):140-8. doi: 10.3109/0284186X.2015.1049290. Epub 2015 Jul 10. PMID 26161618